CLINICAL TRIAL: NCT00743743
Title: Randomized, Placebo-controlled Clinical Trial of Resveratrol Supplement Effects on Cognition, Function and Behavior in Patients With Mild-to-moderate Alzheimer's Disease
Brief Title: Pilot Study of the Effects of Resveratrol Supplement in Mild-to-moderate Alzheimer's Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: PI has left institution
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Resveratrol2008
Record Dates: First submitted 2008-08-27; First posted 2008-08-29 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Alzheimer Disease
Keywords: dementia; Alzheimer disease; cognition; function; behavior; treatment
MeSH Terms: conditions — Alzheimer Disease; Dementia; Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): receive 1 Longevinex brand capsule daily containing 215 mg of resveratrol active ingredient
  Interventions: Dietary Supplement: Longevinex brand resveratrol supplement
- 2 (Placebo Comparator): Receive 1 capsule daily for 52 weeks containing placebo for comparison to experimental arm
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Longevinex brand resveratrol supplement — 1 capsule daily for 52 weeks containing 215 mg of resveratrol active ingredient
  Other Names: Longevinex brand to manufacture the active capsules and placebo capsules for the purposes of this study.
  Arms: 1
Dietary Supplement: placebo — 1 capsule of placebo daily for 52 weeks
  Other Names: Longevinex brand to manufacture placebo capsules to be identical to active agent capsules
  Arms: 2

SUMMARY:
Objective: To determine the effects of resveratrol extract given in a 215 mg dose in a daily supplement currently available over the counter, on cognitive and global functioning in patients with mild to moderate AD on standard therapy.

DETAILED DESCRIPTION:
Background: Many animal and in vitro studies have shown that resveratrol, a naturally occurring polyphenol found in red wine, can increase cognition, reduce neural degeneration, promote clearance of amyloid-beta peptides, and alter aging mechanisms. Therefore, resveratrol may reduce the symptoms of Alzheimer's disease (AD) and possibly its pathology. Objective: A pilot study to determine the effects of resveratrol on cognitive, behavioral and global functioning in patients with mild-to-moderate AD on standard therapy. Design: Randomized, double-blind, placebo-controlled clinical trial. Participants: 50 patients with mild-moderate Alzheimer's disease (AD) defined as a Mini-Mental State Exam (MMSE) between 10-27 will be enrolled in the study. Patients must have an established diagnosis of AD by NINCDS diagnostic criteria, be on stable dose of cognitive enhancing medications (cholinesterase inhibitor and/or NMDA receptor antagonist) Screening/Enrollment: Institutional Review Board approval will be obtained. The chart review and the enrollment discussion will be carried out by a non-physician member of the research team. Participants will be screened and randomized until a total of 50 eligible patients, 25 in each arm are obtained.

ELIGIBILITY:
Inclusion Criteria

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male or female subject with a clinical diagnosis of probable Alzheimer's disease in accordance with NINCDS-ADRDA criteria (Appendix 2).
2. Subject has mild to moderate Alzheimer's disease as defined by a MMSE score 10 to 27 inclusive at Screening.
3. Hachinski Ischemia Score ≤ at Screening (See Appendix 3).
4. Age ≥50 and ≤90 years.
5. At least 6 months of ongoing acetylcholinesterase inhibitor therapy for Alzheimer's disease, with stable dosing for at least the last 2 months (and with no intent to change for the duration of the study).
6. Current use of medication is in accordance with the criteria listed in Table 2 (Permitted Medications, Section 8.1 ).
7. Female subjects must be post-menopausal (i.e. >24 weeks without menstrual period), surgically sterile, or agree to use adequate method of contraception for the duration of the study. Female subjects who are pre-menopausal or who have been post-menopausal for <2 years must undertake pregnancy testing (urine test) at Visit 1, which must be negative.
8. Brain CT or MRI scan performed within the past 12 months or at Screening, showing no evidence of any other potential cause of dementia other than Alzheimer's disease.
9. Neurological exam without focal changes (excluding changes attributable to AD or peripheral trauma).
10. Subject has the ability to comply with procedures for cognitive and other testing.
11. Subject lives with (or has substantial periods of contact with) a regular caregiver who is willing to attend all visits, oversee the subject's compliance with protocol-specified procedures and study medication, and report on subject's status.
12. Subject has provided full written informed consent prior to the performance of any protocol-specified procedure; or if unable to provide informed consent due to cognitive status, full written informed consent on behalf of the subject has been provided by a legally acceptable representative.
13. Caregiver has provided full written informed consent on his/her own behalf prior to the performance of any protocol-specified procedure.

Exclusion Criteria

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Diagnosis of possible, probably, or definite vascular dementia in accordance with NINDS-AIREN criteria (Appendix 4).
2. History or evidence of any other CNS disorder that could be interpreted as a cause of dementia; e.g. cerebrovascular disease (stroke, hemorrhage), structural abnormality, epilepsy, infectious or inflammatory/demyelinating CNS conditions, Parkinson's disease.
3. Evidence of the following disorders: current vitamin B12 deficiency, positive syphilis serology, or active thyroid dysfunction (particularly that suggestive of hypothyroidism), including abnormally high or low serum levels of thyroid stimulating hormone (TSH) that is clinically significant in the opinion of the investigator.
4. History of Type 1 diabetes mellitus or secondary diabetes mellitus.
5. Type 2 diabetes mellitus where the subject is being treated with insulin, a PPARγ agonist, or an insulin secretagogue (e.g. a sulfonylurea or glitinide).
6. Any patient with an HbA1c≥8.5%. (See Section 6.3.8.4 for Safety Measures for Enrolled Subjects with Type 2 Diabetes Mellitus.)
7. History or clinical/investigational evidence of congestive heart failure defined by the New York Heart Association criteria (Class I to IV cardiac status; Appendix 5).
8. History of cardiovascular event within the last 6 months (i.e. intervention, percutaneous coronary intervention, vascular surgery, acute coronary syndrome [non Q-wave myocardial infarction, Q-wave myocardial infarction, unstable angina] or significant arrhythmia; or major intervention (e.g. cardiac surgery or angiography plus stenting) scheduled).
9. History of significant psychiatric illness such as schizophrenia or bipolar affective disorder that in the opinion of the Investigator would interfere with participation in the study, major depressive disorder (according to DSM-IV) in the past year, or current active depression requiring treatment.
10. History or presence of gastro-intestinal, hepatic, or renal disease or other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs, ,or any other clinically relevant abnormality, medical or psychiatric condition, which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study.
11. Clinically significant peripheral edema at the time of screening.
12. Current or recent drug or alcohol abuse or dependence (defined by DSM-IV criteria for substance-related disorders), or recent or remote history of the same if that could be a contributing factor to the dementia.
13. Systolic blood pressure >165 or <90 mmHg or diastolic blood pressure >95 or <60 mmHg at the time of screening.
14. Clinically significant anemia (i.e. hemoglobin >11 g/dL for males or <10 g/dL for females) or presence of hemoglobinopathies which would prevent accurate assessment of HbA1c.
15. Abnormal kidney function tests (>1.5 times the upper limit of normal (ULN)).
16. ALT, AST, or alkaline phosphatase values >2.5 times the ULN, total bilirubin values >1.5 times the ULN, or history of severe hepatobiliary disease (e.g. hepatitis B or C, or cirrhosis, Child-Pugh Class B/C).
17. History of bone marrow transplant.
18. Subject is unable (with assistance, if appropriate) to take study medication as prescribed throughout the study or is at risk of non-compliance with study medication or procedures.
19. Subject is an immediate family member or employee of the participating Investigator, of any of the participating site staff.

    -

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
cognition | 52 weeks

SECONDARY OUTCOMES:
function | 52 weeks
behavior | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diana R Kerwin, MD, Principal Investigator — Medical College of Wisconsin